CLINICAL TRIAL: NCT05941390
Title: Using Virtual Reality (VR) Technology in Gynecological Procedures
Brief Title: Using Virtual Reality (VR) Technology in Gynecological and Obstetrics Procedures
Acronym: VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0125-22-AAA
Record Dates: First submitted 2023-06-05; First posted 2023-07-12 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-06

CONDITIONS: Virtual Reality; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): patients undergoing one of the procedures without using VR device
- VR without sound (Active Comparator): patients undergoing one of the procedures using VR device without sound
  Interventions: Device: VR without positive psychology
- VR with sound (Active Comparator): patients undergoing one of the procedures using VR device with sound
  Interventions: Device: VR with positive psychology

INTERVENTIONS:
Device: VR without positive psychology — Using VR goggles showing relaxing short videos without sound
  Arms: VR without sound
Device: VR with positive psychology — Using VR goggles showing relaxing short videos with positive psychological messages
  Arms: VR with sound

SUMMARY:
A randomized control trial will be conducted in Assuta Ashdod hospital, in the department of obstetrics and gynecology. Pregnant and non pregnant women, undergoing one of the procedures (external cephalic version,amniocentesis or hysteroscopy), will be approached. All willing patients meeting the criteria will sign an informed consent form will.

After signing informed consent patients will be randomly allocated into three groups:1) control (no use of VR). 2) use of VR googles without positive psychology. 3) use of VR googles with positive psychology.

Before and after the procedure each group will answer pain and anxiety questionnaires. In addition, following, following each procedure, salivary cortisol levels will be measured.

ELIGIBILITY:
Inclusion Criteria:

* ECV- single tone, breech presentation,gestional age 35-40,unknown drug allergy
* amniocintesis -single tone,gestional age 16-24 week,
* hysteroscopy-women age 18-60 , diagnostic procedure,

Exclusion Criteria:

* ECV-previous cesarian section, contruction,low known plt count ,premature rupture of membrane
* amniocintesis- Known fetal malformations, amnionitis
* hysteroscopy-pregnancy, PID

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
stress cortisol saliva level | up to 5 minutes after the procedure
  each arm after the procedure will be mesured stress cortisol level in saliva

SECONDARY OUTCOMES:
pain levels | up to 5 minutes after
  each arm after the procedure will fill pain questioner. pain questioners using visual analog score. 0- to 10, while 0 is no pain at all, 10 is the worse pain ever felt.the patients will fill the questioner before and after the procedures.
anxiety levels | up to 5 minutes after
  each arm after the procedure will fill anxiety questioner. anxiety questioner using the short depression , anxiety and stress scale (DASS-21). the patients will fill the questioners before and after the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Noa glick fishman, MD, Principal Investigator — Assuta Ashdod

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koyyalamudi V, Sidhu G, Cornett EM, Nguyen V, Labrie-Brown C, Fox CJ, Kaye AD. New Labor Pain Treatment Options. Curr Pain Headache Rep. 2016 Feb;20(2):11. doi: 10.1007/s11916-016-0543-2. PMID 26780039
- [Background] Woolf CJ. What is this thing called pain? J Clin Invest. 2010 Nov;120(11):3742-4. doi: 10.1172/JCI45178. Epub 2010 Nov 1. PMID 21041955
- [Background] Frey DP, Bauer ME, Bell CL, Low LK, Hassett AL, Cassidy RB, Boyer KD, Sharar SR. Virtual Reality Analgesia in Labor: The VRAIL Pilot Study-A Preliminary Randomized Controlled Trial Suggesting Benefit of Immersive Virtual Reality Analgesia in Unmedicated Laboring Women. Anesth Analg. 2019 Jun;128(6):e93-e96. doi: 10.1213/ANE.0000000000003649. PMID 31094789
- [Background] Wong MS, Spiegel BMR, Gregory KD. Virtual Reality Reduces Pain in Laboring Women: A Randomized Controlled Trial. Am J Perinatol. 2021 Aug;38(S 01):e167-e172. doi: 10.1055/s-0040-1708851. Epub 2020 Jun 2. PMID 32485759